CLINICAL TRIAL: NCT02312830
Title: Belgian Cross-sectional Allogeneic Transplant Survivor Study
Acronym: BE-C@TS
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57284
Record Dates: First submitted 2014-10-15; First posted 2014-12-09 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hematopoietic Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation, Allogeneic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
With the increasing successful use of allogeneic hematopoietic stem cell transplantation (HSCT) to cure advanced hematological disease, it becomes essential to evaluate the long-term effects of such a drastic treatment.

This study investigates the prevalence of several demographic, psychosocial and behavioral aspects of survivorship after an allogeneic transplantation. Income, return to work, social isolation, pain, medication adherence, influenza vaccination status, alcohol use, smoking habits, drug use, healthy diet, prevention of UV exposure, physical activity, functional status/Quality of life (QoL), couple life/sexual function, depression, anxiety, spirituality and resilience will be studied.

DETAILED DESCRIPTION:
This is a cross sectional study, where participants are interviewed and fill in a self reported survey. The interview and survey are only taken once. It is non interventional because the patients only give us extra information, which is not usually recorded in our medical records.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in Dutch
* Age above 18 years at time of transplant
* Transplanted in UZ Leuven between 1992 and 2012 with an allogeneic donor (i.e. being at least 2 years post-Tx)
* Presenting for a periodic health check in UZLEUVEN from November 15th, 2014 to November 15th 2016
* Willing to provide oral and written consent

Exclusion Criteria:

* Unable to communicate fluently in Dutch
* Presenting with major visual, hearing, cognitive or psychiatric conditions precluding participation
* Presenting with relapse or other major illness, with less than 6 months expected survival
* Hospitalized for a life-threatening condition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients transplanted in UZ Leuven between 1992 and 2012 with an allogeneic donor (i.e. being at least 2 years post-Tx) - Hematopoietic Stem Cell Transplantation, presenting for a standard medical check up
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
composite outcome: prevalence of several demographic, psychosocial and behavioral aspects of survivorship after an allogeneic transplantation | The interview/survey will happen once per patient and will be offered to all transplant survivors (minimum 2 years post transplant) coming to the clinic between Nov 2014-Nov 2016. No follow up included.
  This is a cross sectional study, assessing several aspects of survivorship with multiple validated questionnaires (EQ5D, PHQ9, GAD, SFQ, etc). These questionnaires are only taken once in all survivors approached for the study.